CLINICAL TRIAL: NCT02189499
Title: Amaranth Endovascular Study of a Drug-Eluting Bioresorbable Coronary Scaffold
Brief Title: Feasibility Study of the Amaranth Medical FORTITUDE Bioresorbable Drug-Eluting Coronary Stent
Acronym: MEND II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amaranth Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0170
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Stents; Angioplasty; Coronary Vessels; Coronary Artery Disease; Angina Pectoris; Myocardial Ischemia; Myocardial Infarction; Myocardial Revascularization
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coronary Scaffold Implantation (Experimental): AmM FORTITUDE Bioresorbable Drug-Eluting Coronary Scaffold
  Interventions: Device: AmM FORTITUDE Bioresorbable Drug-Eluting Coronary Scaffold

INTERVENTIONS:
Device: AmM FORTITUDE Bioresorbable Drug-Eluting Coronary Scaffold — Placement of the investigational device into the diseased coronary artery to eliminate the vascular stenosis.
  Other Names: Coronary stent

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of a new coronary artery stent for treating blockages in the arteries supplying blood to the heart muscle. The Amaranth FORTITUDE scaffold releases a drug (sirolimus) to reduce the likelihood of the treated blood vessel developing a new blockage. In addition, the scaffold dissolves away over time, leaving no permanent implant after the blood vessel has healed. This study will will be the first evaluation of this stent in humans.

DETAILED DESCRIPTION:
The objective of this first-in-man study is to evaluate the safety and feasibility of the AmM FORTITUDE Bioresorbable Drug-Eluting Coronary Scaffold for use in the treatment of single, de novo, stenotic native coronary artery lesions in patients undergoing elective percutaneous coronary intervention. The scaffold is a single-use device comprised of a balloon-expandable, intracoronary drug coated scaffold pre-mounted on a rapid-exchange delivery catheter. The scaffold is made of Poly-L-Lactide (PLLA) and is coated with a polymer-antiproliferative drug (sirolimus) matrix. The scaffold provides mechanical support similar to a metallic stent to the vessel while it is healing, and then gradually breaks down over time leaving no permanent implant in the treated vessel.

The study design is a prospective, non-randomized, feasibility trial. It will enroll a maximum of 50 patients from multiple investigational centers in Columbia. Eligible patients who are at least 18 years of age diagnosed with symptomatic ischemic disease due to a discrete, single, de novo, stenotic lesion in native coronary artery will be asked to participate in this study. After treatment with the investigational device, subjects will be followed for five years. Safety of the device will be evaluated using the incidence of target vessel failure during the follow-up period. Efficacy will be assessed using the in-scaffold late lumen loss measured by quantitative coronary angiography at nine months.

ELIGIBILITY:
Inclusion Criteria:

General

1. Subject is ≥ 18 years of age and < 85 years of age.
2. Subject agrees not to participate in any other investigational device or drug study for a period of two years following the index procedure. Questionnaire-based studies, or other studies that are non-invasive and do not require investigational devices or medications are allowed.
3. Subject (or their legally authorized representative) provides written informed consent prior to any study-related procedure, using the form approved by the local Ethics Committee.
4. Subject has:

   1. evidence of myocardial ischemia (e.g., stable angina [Canadian Cardiovascular Society 1, 2, 3, or 4] or unstable angina [Braunwald Class 1-3, B-C], or silent ischemia with supporting imaging studies [ETT, SPECT, stress echocardiography, or Cardiac CT]), or
   2. low or intermediate risk NSTEMI, or
   3. evidence of myocardial ischemia in a coronary territory previously affected by STEMI as long as the lesion fulfills the angiographic inclusion criteria and the intervention performed ≥ 6 months following the clinical event.
5. Subject is an acceptable candidate for coronary artery bypass graft (CABG) surgery.
6. Patient agrees to complete all protocol required follow-up visits, including angiograms and OCT exams.
7. Percutaneous interventions for lesions in a non-target vessel are allowed if done ≥ 30 days prior to or planned to be done ≥ 9 months after the index procedure.
8. Percutaneous interventions for lesions in the target vessel are allowed if done ≥ 6 months prior to or planned to be done ≥ 9 months after the index procedure.

Angiographic

1. Patient indicated for elective stenting of a single, de novo, stenotic lesion in a native coronary artery.
2. Target lesion must measure ≤ 14 mm in length by on-line QCA.
3. Lesion must be located in a native coronary artery with a diameter (average of distal and proximal to lesion by IVUS) of 2.5 mm to 3.7 mm.
4. Target lesion must be in a major artery or branch with a visually estimated diameter stenosis of ≥ 50% and < 100% with a Thrombolysis in Myocardial Infarction (TIMI) flow of ≥ 1.

Exclusion Criteria:

General

1. Patient has known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel, prasugrel, and ticagrelor), poly (L-lactide), platinum-iridium, or contrast sensitivity that cannot be adequately pre-medicated.
2. Patient has evolving ST segment elevation myocardial infarction (STEMI).
3. Patient has current unstable arrhythmias.
4. Patient has a left ventricular ejection fraction (LVEF) < 30%.
5. Patient has received a heart transplant or any other organ transplant, or is on a waiting list for any organ transplant.
6. Patient has any previous stent placements ≤ 15 mm (proximal or distal) of the target lesion.
7. Patient is receiving or scheduled to receive chemotherapy for malignancy ≤ 30 days prior to or after the index procedure.
8. Patient is receiving immunosuppressant therapy and/or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus, rheumatoid arthritis, severe asthma requiring immunosuppressive medication, etc.).
9. Patient is receiving or scheduled to receive chronic anticoagulation therapy (e.g., heparin, Coumadin) that cannot be stopped and restarted according to local hospital standard procedures.
10. Elective surgery is planned ≤ 9 months after the index procedure that will require discontinuation of anti-platelet medications.
11. Patient has a platelet count < 100,000 cells/mm^3 or > 700,000 cells/mm^3, a WBC of < 3,000 cells/mm^3, or documented or suspected liver disease (including laboratory evidence of hepatitis).
12. Patient has known renal insufficiency (e.g., eGFR < 60 ml/kg/m^2 or serum creatinine level of > 2.5 mg/dL, or subject on dialysis).
13. Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
14. Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) ≤ 6 months prior to the index procedure.
15. Patient has had a significant GI or urinary bleed ≤ 6 months prior to the index procedure.
16. Patient has extensive peripheral vessel disease that precludes safe introducer sheath insertion.
17. Patient has received brachytherapy in any epicardial vessel (including side branches).
18. Pregnant or nursing subjects and those who plan pregnancy ≤ 2 years following index procedure. (Note: Female subjects of child-bearing potential must have a negative pregnancy test ≤ 28 days prior to the index procedure and agree to use contraception for 2 years.)
19. Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy (i.e., ≤ 1 year).
20. Subject belongs to a vulnerable population (per investigator's judgment, e.g., subordinate hospital staff, mentally deficient, or unable to read or write).

Angiographic Exclusion

1. Target lesion meets any of the following criteria:

   1. Aorto-ostial location (within ≤ 3 mm of aorta junction).
   2. Left Main location.
   3. Located ≤ 3 mm of the origin of the left anterior descending (LAD) or left coronary circumflex (LCX).
   4. Located within an arterial or saphenous vein graft or distal to a diseased (defined as vessel irregularity per angiogram and > 20% stenosed lesion, by visual estimation) arterial or saphenous vein graft.
   5. Lesion involving a bifurcation > 2 mm in diameter and ostial lesion > 40% stenosed by visual estimation or side branch requiring predilatation.
   6. Total occlusion (TIMI flow 0) prior to wire crossing.
   7. Excessive tortuosity (≥ two 45° angles), or extreme angulation (≥ 90°) proximal to or within the target lesion.
   8. Restenotic from previous intervention.
   9. Moderate to severe superficial calcification (defined as calcium arch > 120°) proximal to or within the target lesion.
2. Target lesion involves myocardial bridge.
3. Target vessel contains visible thrombus as indicated in the angiographic images.
4. Another clinically significant lesion is located in the same major epicardial vessel as the target lesion (including side branches).
5. Inadequate pre-dilation of the target lesion (residual stenosis > 40% by visual assessment).
6. Patient has a high probability that the use of other ancillary devices such as atherectomy or cutting balloon will be required at the time of index procedure for treatment of the target vessel.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of target vessel failure | 9 months
  Defined as the composite rate of cardiac death (using the Academic Research Consortium [ARC] definition), target vessel myocardial infarction (using the Third Universal Definition of MI), or clinically indicated target lesion revascularization (using the ARC definition).
In-scaffold late lumen loss | 9 months
  Defined as the amount of vessel lumen diameter (in mm) lost/gained at the time of follow-up compared to the immediate post-treatment result, as measured by quantitative coronary angiography (QCA). The assessment is made within the segment of vessel including the scaffold.

SECONDARY OUTCOMES:
Clinical device success | intraoperative
  Defined as successful delivery and deployment of the investigational scaffold at the intended target lesion with attainment of a final residual stenosis of < 50% of the target lesion by quantitative coronary angiography (QCA) after the index procedure.
Clinical procedure success | Participants will be followed for the duration of their hospital stay, an expected average of 1-2 days
  Defined as successful delivery and deployment of the investigational scaffold at the intended target lesion, with attainment of a final residual stenosis of < 50% of the target lesion by quantitative coronary angiography (QCA) using any adjunctive device, without the occurrence of major adverse clinical events (cardiac death, target vessel myocardial infarction, or clinically indicated target lesion revascularization) during the duration of the subject's hospital stay (an average of 1-2 days).

OTHER OUTCOMES:
In-segment/in-scaffold late lumen loss | 9 months and 2 years
  Defined as the amount of vessel lumen diameter (in mm) lost/gained at the time of follow-up compared to the immediate post-treatment result, as measured by quantitative coronary angiography; the assessment is made both within the scaffold itself ("in-scaffold") and within the segment of vessel including the scaffold and 5 mm proximal and distal to the scaffold ("in-segment").
In-scaffold percent volume obstruction | 9 months and 2 years
  Defined as the difference between the volume enclosed within the scaffold and the corresponding vessel lumen, expressed as a percentage of the scaffold volume at the time of follow-up, measured using optical coherence tomography (OCT)
Stent thrombosis | Hospital discharge, 30 days, 9 months, and 2 years
  Defined using the ARC "definite" or "probable" stent thrombosis definitions.
In-scaffold/in-segment binary restenosis rate | 9 months and 2 years
  Defined as the percentage of treated coronary lesions with a residual diameter stenosis over 50% at the time of follow-up, as measured by quantitative coronary angiography (QCA). The assessments are made both within the scaffold itself ("in-scaffold") and within the segment of vessel including the scaffold and 5 mm proximal and distal to the scaffold ("in-segment").
Incomplete scaffold strut apposition to the vessel wall | 9 months and 2 years
  Defined as the number (or percentage) of scaffold struts not in direct contact with the vessel wall, either persisting from the implantation of the scaffold or newly occurring after the time of scaffold implantation, assessed at follow-up using OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Granada, MD, Principal Investigator — Skirball Center for Cardiovascular Research, Columbia University Medical Center
Locations (4):
- Colombia (4):
  - Clinica de Marly, Bogotá
  - Instituto del Corazon, Bucaramanga
  - Angiografia De Occidente S.A., Cali
  - EMMSA Clinica Especializada, Medellín

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Granada JF. The Amaranth PLLA based bioresorbable scaffold (ABRS): Experimental and early human results. TCT presentation 2013.
- [Background] Granada JF. BRS with clinical data III, Amaranth: Differentiating features and clinical update. TCT presentation 2014.